CLINICAL TRIAL: NCT04321655
Title: Reduce Pain and Improve Quality of Life in Patient With Knee Osteoarthritis by Light, Sound and Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/IEC/110P; U1111-1248-7814 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-17; First posted 2020-03-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; uphill; incline walking; degeneration; laser therapy; ultrasound; tDCS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Intensity LASER Therapy group (HILT) (Experimental): Forty patients with chronic KOA in HILT group will received Class IV LASER therapy. A Class IV LASER emits power more than 500 milliwatt (mW) .
  Interventions: Other: High Intensity LASER Therapy (HILT)
- Ibuprofen gel phonophoresis (IGP) group (Experimental): Patients with chronic KOA in ibuprofen gel phonophoresis (IGP) group will administered with continuous ultrasound set at a frequency of 1 megahertz (MHz) and an intensity of 1 W/cm2 was applied on a circular basis.
  Interventions: Other: Ibuprofen Gel Phonophoresis (IGP)
- Transcranial direct current stimulation (tDCS) group (Experimental): Fourty patients with chronic KOA will receive structured tDCS (MA-tDCS, Walnut-Medical, Johnstown, PA) treatment. Two pair of sponge electrodes soaked with saline and fixed to head with elastic bands. The transcranial direct current stimulation will be applied by a constant current device with an intensity of 2mA
  Interventions: Other: Transcranial Direct Current Stimulation (tDCS)
- Conventional physiotherapy group (CPT) (Active Comparator): Individual with chronic KOA will be educated on how to do the set of exercises correctly at their home during the first session. All the groups will receive the same, standardized exercise protocol for KOA which consisted of nine exercises including muscle strengthening and flexibility training.
  Interventions: Other: Conventional Physiotherapy (CPT)

INTERVENTIONS:
Other: High Intensity LASER Therapy (HILT) — The total energy will be delivered to the patient during one session will be 1,250 J through three phases of treatment.
  1. Initial phase (710 and 810 mJ (millijoule)/cm2 for a total of 500 J)
  2. Intermediate phase (handpiece will be applied on the joint line just proximal to the medial and lateral tibial condyles with 25 J, a fluency of 610 mJ/cm2, and a time of 14 s for each point and a total of 250 J)
  3. Final phase (same as the initial phase (500 J) except that scanning will be slow manual scanning ) The application time for all three phases will be approximately 15 min with the total energy delivered to the patient during one session of 1,250 J
  Arms: High Intensity LASER Therapy group (HILT)
Other: Ibuprofen Gel Phonophoresis (IGP) — Continuous ultrasound set at a frequency of 1 MHz and an intensity of 1 W/cm2 was applied on a circular basis. (8 min/ one session each day for 3 days/week for 8 weeks).
  Arms: Ibuprofen gel phonophoresis (IGP) group
Other: Transcranial Direct Current Stimulation (tDCS) — Anode electrode -C3/C4 (contralateral side of the most affected knee), Cathode electrode- contralateral supraorbital area. (2 mA intensity for 20 minutes, one session/day for 3 days/week for 8 weeks)
  Arms: Transcranial direct current stimulation (tDCS) group
Other: Conventional Physiotherapy (CPT) — 1. Warm-up exercises: Walking at the usual speed on a flat surface for 10 min ( 3sets X10 Reps X 3 min rest in between)
  2. Hamstring and calf gentle stretches. ( 3sets X10 Reps X 3 min rest in between)
  3. Straight leg raise (SLR) ( 3sets X10 Reps X 3 min rest in between)
  4. Quadriceps setting ( 3sets X10 Reps X 3 min rest in between)
  5. Pillow squeeze ( 3sets X10 Reps X 3 min rest in between)
  6. Heel raise ( 3sets X10 Reps X 3 min rest in between)
  7. One leg balance ( 3sets X10 Reps X 3 min rest in between)
  8. Step ups ( 3sets X10 Reps X 3 min rest in between)
  9. Quadriceps strengthening exercises ( 3sets X10 Reps X 3 min rest in between)
  Arms: Conventional physiotherapy group (CPT)

SUMMARY:
Patients affected with osteoarthritis knee have associated with pain and inflammation of the joint capsule, impaired muscular stabilization, decrease range of motion and functional disability. Laser therapy, phonophoresis, transcranial direct current stimulation (tDCS) and conventional physiotherapy exercises has innumerable benefits to the patients with knee osteoarthritis (KOA).However, it is still not clear which treatment is effective among them in rehabilitating the patients with chronic knee osteoarthritis (KOA). Aim is to establish the benefits of High intensity Laser therapy, phonophoresis, tDCS and conventional physiotherapy in the treatment of patient with chronic KOA living in the hilly terrain. A total of 160 patients with chronic KOA will be recruited by the simple random sampling (random number generator) to participate in randomized, double blind randomized controlled, study. Recruited patients with chronic KOA will be randomly divided into four groups, high intensity-laser therapy (HILT) group, ibuprofen gel phonophoresis (IGP) group, transcranial direct current stimulation (tDCS) group and conventional physiotherapy (CPT) group. Duration of the treatment will be 8 minutes in one session/knee joint for HILT and IGP and 30 minutes in one session for tDCS each day for 3 days/week for 8 weeks. Thus, each patient with chronic KOA will receive 24 sessions in total. The Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC), Digitalized pain pressure algometer (ALGO-DS-01) and 36-Item Short Form Health Survey (SF-36) questionnaire are the outcome measures will be recorded at baseline, end of 8-week post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with clinical chronic knee OA according to the diagnostic criteria of American College of Rheumatology (ACR) were included in the study
* Age between 45-70
* Both sex male and female

Exclusion Criteria:

* Unwillingness to participate in the study,
* Recent history (within the last 3 months) of physical therapy to the same joint,
* Recent history (within the last 3 months) of intra-articular procedure (injection and/or lavage) to the knee,
* History of knee surgery/fracture,
* Acute synovitis/arthritis including the infectious conditions,
* Presence of malignancy,
* Pregnancy
* Taking pain relief medications
* Any metal implants near the site of stimulation

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-08-02 (Estimated)

PRIMARY OUTCOMES:
Digitalized pain pressure algometer | Changes will be measured at baseline and end of 8 week intervention
  Pain intensity will be measured using calibrated digitalized pain pressure algometer (ALGO-DS-01) in patients with KOA. Sensor digital algometer is force gauge with computer size which is highly accurate. The ALGO-DS-01 is chosen for the assessment of pain for Mechanical sacroiliac joint dysfunction, which is a reliable and valid tool for assessing sacroiliac joint dysfunction. The inter rater reliability of pressure pain algometer was demonstrated to be moderate to good reliability with interclass correlation coefficient (ICC) of (0.62-0.84)
Western Ontario and Mc Master Universities Osteoarthritis Index | Changes will be measured at baseline and end of 8 week intervention
  The Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC) will be was used to evaluate the disease-specific self-reported symptoms of OA.48 This form is comprised of 24 questions in three categories including pain (5 questions), stiffness (2 questions), and physical function (17 questions). These 24 items are presented in a five-point Likert (0-4) scale, where higher scores indicate the higher intensity of the related symptom. The minimal clinical important difference of WOMAC at 2 month of intervention is found to be, 14.1 The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
36-Item Short Form Health Survey | Changes will be measured at baseline and end of 8 week intervention
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life (QoL). The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). SF-36 is used to assess QoL in patient with KOA.
  The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh K Srivastav, MPT, Principal Investigator — Maharishi Markandeshwar Medical College and Hospital; Asir J Samuel, MPT, Ph.D, Study Chair — Maharishi Markandeshwar Medical College and Hospital; Vipin Saini, Ph.D, Study Director — Maharishi Markandeshwar Medical College and Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WJ, Bennell KL, Hodges PW, Hinman RS, Young CL, Buscemi V, Liston MB, Schabrun SM. Addition of transcranial direct current stimulation to quadriceps strengthening exercise in knee osteoarthritis: A pilot randomised controlled trial. PLoS One. 2017 Jun 30;12(6):e0180328. doi: 10.1371/journal.pone.0180328. eCollection 2017. PMID 28665989
- [Result] Stiglic-Rogoznica N, Stamenkovic D, Frlan-Vrgoc L, Avancini-Dobrovic V, Vrbanic TS. Analgesic effect of high intensity laser therapy in knee osteoarthritis. Coll Antropol. 2011 Sep;35 Suppl 2:183-5. PMID 22220431
- [Result] Coskun Benlidayi I, Gokcen N, Basaran S. Comparative short-term effectiveness of ibuprofen gel and cream phonophoresis in patients with knee osteoarthritis. Rheumatol Int. 2018 Oct;38(10):1927-1932. doi: 10.1007/s00296-018-4099-9. Epub 2018 Jul 12. PMID 30003324
- [Result] Srivastav AK, Sharma N, Samuel AJ. tDCS combined with cognitive training in a patient with chronic traumatic head injury. Neurophysiol Clin. 2020 Apr;50(2):133-134. doi: 10.1016/j.neucli.2020.02.004. Epub 2020 Mar 5. No abstract available. PMID 32147282